CLINICAL TRIAL: NCT07133776
Title: A Multicenter, Single-Arm, Prospective Clinical Study to Evaluate the Efficacy and Safety of PD-1 Inhibitor Combined With Tenofovir, Chidamide, and Lenalidomide in the Treatment of EBV-Associated Diseases
Brief Title: Application of PD-1 Inhibitors Combined With Tenofovir, Chidamide and Lenalidomide in the Treatment of EBV-associated Diseases.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL294-01
Record Dates: First submitted 2025-07-30; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Epstein-Barr Virus (EBV) Infection; PD-1 Inhibitor; Tenofovir; Chidamide; Lenalidomide
Keywords: Epstein-Barr Virus (EBV) infection; PD-1 Inhibitor; tenofovir; Chidamide; lenalidomide
MeSH Terms: conditions — Epstein-Barr Virus Infections; Infections | interventions — Tenofovir; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluate efficacy and safety of multi-drug therapy in EBV infectious diseases. (Experimental): To investigate the therapeutic effect of PD-1 inhibitor combined with tenofovir, chidamide, and lenalidomide in EBV infectious diseases, and to evaluate its safety and clinical benefit in this patient population.
  Interventions: Drug: PD-1 Inhibitor Combined with Tenofovir, Chidamide, and Lenalidomide for the Treatment of EBV Infectious Diseases.

INTERVENTIONS:
Drug: PD-1 Inhibitor Combined with Tenofovir, Chidamide, and Lenalidomide for the Treatment of EBV Infectious Diseases. — This study involves a four-drug combination regimen consisting of a PD-1 inhibitor, tenofovir, chidamide, and lenalidomide for the treatment of EBV Infectious diseases, aiming to inhibit viral replication and restore immune function through multiple mechanisms. The intervention includes not only pharmacological treatment but also pre-treatment assessments (such as EBV-DNA load, immune status, cardiac and renal function), efficacy monitoring during treatment (e.g., ORR, changes in EBV-DNA), and post-treatment follow-up for safety and survival outcomes (including OS, PFS, and adverse events), in order to comprehensively evaluate the clinical value and feasibility of this combination therapy.

SUMMARY:
Currently, treatment options for Epstein-Barr virus (EBV) infection are limited, with unsatisfactory efficacy and no established standard therapy. Therefore, our center is conducting a prospective, multicenter, single-arm clinical trial to evaluate the efficacy and safety of PD-1 inhibitor in combination with tenofovir, chidamide, and lenalidomide in patients with EBV infectious diseases, aiming to provide a more effective and safer therapeutic option for EBV infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with EBV infectious diseases, including infectious mononucleosis, chronic active EBV infection, or other EBV infectious diseases;
2. EBV DNA ≥ 10⁴ copies/mL in whole blood or plasma;
3. Age ≤ 75 years with ECOG performance status ≤ 2;
4. Estimated life expectancy over 3 months;
5. Patients must be able to undergo follow-up. They should understand the nature of their disease and voluntarily agree to participate in this study for treatment and follow-up.

Exclusion Criteria:

1. Patients with impaired liver or kidney function, specifically defined as serum direct bilirubin, indirect bilirubin, and/or ALT, AST, or serum creatinine >2 times the upper limit of normal (ULN), unless such abnormalities are attributed to lymphoma;
2. Patients with bone marrow failure, defined as absolute neutrophil count (ANC) <1.5×10⁹/L or platelets <75×10⁹/L;
3. Patients who have experienced grade III or higher neurotoxicity within the past 2 weeks;
4. Patients with chronic heart failure classified as NYHA class III or IV, or left ventricular ejection fraction (LVEF) <50%, or those with a history of the following cardiac events within the past 6 months: acute coronary syndrome, acute heart failure (NYHA class III or IV), or significant ventricular arrhythmias (sustained ventricular tachycardia, ventricular fibrillation, or resuscitated sudden cardiac arrest);
5. Patients with AIDS, syphilis, or active hepatitis B (HBV DNA >1×10⁴ copies/mL) or hepatitis C infection;
6. Patients with coexisting hematologic disorders (e.g., hemophilia, myelofibrosis) deemed unsuitable for inclusion by the investigator;
7. Patients with severe concurrent infections;
8. Patients who have undergone grade II or higher surgery within 3 weeks prior to treatment;
9. Patients with substance abuse, medical, psychological, or social conditions that may interfere with study participation or the evaluation of study outcomes;
10. Patients deemed unsuitable for enrollment by the investigator;
11. Patients with known hypersensitivity to components of the investigational drug.

Ages: 0 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR), including Complete Response (CR) and Partial Response (PR), based on EBV-DNA levels. | After 3 months of treatment according to the study protocol, a comprehensive efficacy assessment will be conducted. Patients achieving CR or PR will continue treatment, while those with SD or PD will be withdrawn from the study.

SECONDARY OUTCOMES:
24-month overall survival rate of EBV-infected diseases. | From first dose until death from any cause (assessed at 24 months）
  Proportion of patients alive at 24 months after initiation of tirelizumab combination therapy.
24-month progression-free survival rate of EBV-infected diseases. | From first dose until first documented progression or death (assessed at 24 months)
  The proportion of patients with no disease progression at 24 months based on EBV DNA results.

IPD SHARING:
Plan to Share IPD: No